CLINICAL TRIAL: NCT00655070
Title: Evaluation of the Effect of T3US on Myocardial Blow Flow in the Hibernating
Brief Title: Effect of Timi3 Ultrasound on Myocardial Blow Flow in the Hibernating Myocardium
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1644-31803-02
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Ischemia
Keywords: Hibernating Myocardium; Blood Flow; Ultrasound; PET imaging
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Timi3 Transthoracic ultrasound — Low frequency ultrasound over the chest using Timi3 ultrasound device

SUMMARY:
The purpose of this study is to evaluate whether the use application of low frequency ultrasound, administered by the Timi3 ultrasound device, increases myocardial blood flow to the heart, in subjects with reduced myocardial blood flow at rest (hibernating myocardium). The primary endpoint of the trial is to assess the increase in myocardial blood flow from baseline to post Timi3 Ultrasound treatment in a hypoperfused region of myocardium. Positron emission tomography (PET) imaging will be used to noninvasively evaluate cardiac blood flow. The hypothesis is that ultrasound increases blood flow in hibernating myocardium.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years
* Must have reversible resting ischemia, resting non-reversible blood flow defect, or stress-induced ischemia.
* Females with childbearing potential must not be pregnant at the time of the study
* Must provide written informed consent

Exclusion Criteria:

* Unable or unwilling to cooperate with study procedures
* Currently enrolled in another clinical study for which the follow-up period is not complete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in myocardial blood flow from baseline to post ultrasound treatment | immediate post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Dae, MD, Principal Investigator — University of California at San Francisco
Locations (1):
- UC San Francisco, San Francisco, California, United States